CLINICAL TRIAL: NCT02077855
Title: Value of Sonographic Diagnosis of Toddler's Fracture of the Tibia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Michael Boettcher, PD Dr. med. Michael Boettcher, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV3964
Record Dates: First submitted 2012-07-09; First posted 2014-03-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Pediatric Fractures
Keywords: Sensitivity and Sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Toddlers fractures

SUMMARY:
This fracture of the distal tibia occurs in 1 to 4 year-old-children. Timely diagnosis is important, because it obviates the need for investigations to archive adequate treatment as well as to prevent unnecessary immobilization. The value of sonographic diagnosis of toddler's fracture has been demonstrated. The aim of the present study is to investigate the reliability and accuracy of sonography in the diagnostic workup of the toddler's fracture.

DETAILED DESCRIPTION:
This fracture of the distal tibia occurs in 1 to 4 year-old-children. The child usually presents with an acute onset of limp or refusal to bear weight on one leg. Toddlers and young children may present with guarding, but may not have swelling or noticeable deformity.

Radiologic signs can be subtle too. In some cases initial radiographs is negative and fractures are diagnosed on follow-up studies by periosteal reaction.

However, timely diagnosis is important, because it obviates the need for investigations to archive adequate treatment as well as to prevent unnecessary immobilization. The value of sonographic diagnosis of toddler's fracture has been demonstrated. In children it is of particular value as it is comfortable and does not involve the use of ionizing radiation.

The aim of the present study is to investigate the reliability and accuracy of sonography in the diagnostic workup of the toddler's fracture.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Suspicion of Toddlers fractures

Exclusion Criteria:

1. Major delay in treatment

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with suspicion of Toddlers fractures.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Sonographic identification of "Toddler's" fractures | 3y
  Comparison of sensitivity and specitivity of sonography and x-ray

SECONDARY OUTCOMES:
US does not cause more discomfort than x-ray | 3y

CONTACTS AND LOCATIONS:
Locations (1):
- UKE Medical School, Hamburg, Germany